CLINICAL TRIAL: NCT01290679
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled Study to Investigate the Efficacy, Safety and Tolerability of TMC435 Versus Placebo as Part of a Treatment Regimen Including Peginterferon α-2a (Pegasys®) and Ribavirin (Copegus®) or Peginterferon α-2b (PegIntron®) and Ribavirin (Rebetol®) in Treatment-naïve, Genotype 1, Hepatitis C-infected Subjects
Brief Title: An Efficacy, Safety, and Tolerability Study of TMC435 in Treatment-naive, Genotype 1 Hepatitis C-infected Participants
Acronym: QUEST-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen R&D Ireland (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR017380; TMC435-TiDP16-C216 (Other: Janssen R&D Ireland); 2010-021174-11 (EudraCT Number)
Record Dates: First submitted 2011-01-07; First posted 2011-02-07 (Estimated); Results first posted 2014-06-13 (Estimated); Last update posted 2014-06-13 (Estimated); Status verified 2014-06

CONDITIONS: Hepatitis C
Keywords: Hepatitis C; TMC435; HCV; Hep C; genotype 1
MeSH Terms: conditions — Hepatitis C | interventions — Simeprevir; peginterferon alfa-2a; peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TMC435 (Experimental): TMC435 150 mg capsule once daily for 12 weeks in addition to peginterferon alfa-2a (Pegasys) or peginterferon alfa-2b (PegIntron) (PegIFN alpha-2a/b) and ribavirin (Copegus or Rebetol) for 24 or 48 weeks
  Interventions: Drug: TMC435; Drug: Peginterferon alpha-2a or Peginterferon alpha-2b (PegIFNα-2a/b); Drug: Ribavirin (RBV)
- Placebo (Placebo Comparator): Placebo 150 mg capsule once daily for 12 weeks in addition peginterferon alfa-2a (Pegasys) or peginterferon alfa-2b (PegIntron) (PegIFN alpha-2a/b) and ribavirin (Copegus or Rebetol) for 48 weeks
  Interventions: Drug: Placebo; Drug: Peginterferon alpha-2a or Peginterferon alpha-2b (PegIFNα-2a/b); Drug: Ribavirin (RBV)

INTERVENTIONS:
Drug: Placebo — 150 mg capsule once daily for 12 weeks in addition to peginterferon alfa-2a or peginterferon alfa-2b and ribavirin for 48 weeks
  Arms: Placebo
Drug: TMC435 — 150 mg capsule once daily for 12 weeks in addition to peginterferon alfa-2a or peginterferon alfa-2b and ribavirin for 24 or 48 weeks
  Arms: TMC435
Drug: Peginterferon alpha-2a or Peginterferon alpha-2b (PegIFNα-2a/b) — One subcutaneous (under the skin) injection of PegIFNα-2a (containing 0.5 mL solution with 180 mcg PegIFNα-2a) OR PegIFNα-2b (0.5 mL from a pre-filled pen) once weekly for up to 48 weeks.
  Other Names: PegIFNα-2a (Pegasys); PegIFNα-2b (PegIntron)
Drug: Ribavirin (RBV) — 200-mg tablets of ribavirin (Copegus or Rebetol) (body-weight adjusted dose) taken orally (by mouth) twice daily for up to 48 weeks.
  Other Names: Copegus; Rebetol

SUMMARY:
The purpose of this study is to investigate the effectiveness and safety of TMC435 compared with placebo in participants who are infected with genotype 1 hepatitis C virus who have never received treatment before. Participants will also receive peginterferon alfa-2a or peginterferon alfa-2b and ribavirin as part of their treatment.

DETAILED DESCRIPTION:
This is a randomized, double-blind (neither physician or participant knows the name of the assigned drug), placebo-controlled study of TMC435 in participants who are infected with genotype 1 hepatitis C virus who have never received treatment for this before. Participants in this study will also receive two other drugs for their infection (either peginterferon alfa-2a (Pegasys®) and ribavirin (Copegus®) or peginterferon alfa-2b (PegIntron®) and ribavirin (Rebetol®). The purpose of the study is to investigate if TMC435 is superior to placebo in reducing hepatitis C virus to an undetectable level 24 weeks after the end of treatment. For the first 12 weeks, participants will take TMC435 or placebo, plus peginterferon and ribavirin. For the next 12 weeks, participants will take peginterferon and ribavirin only. After that, some participants will continue to take peginterferon and ribavirin for up to 24 additional weeks. Other participants will stop taking peginterferon and ribavirin. The study doctor will inform each participant about how to take their study medication and when they should stop taking it. After a participant stops taking study medication, they will continue to come to the doctor's office for study visits until a total of 72 weeks after they enroll in the study. The total duration of the study is 78 weeks (including screening). Participants will be monitored for safety throughout the study. Study assessments at each study visit may include but are not limited to: blood and urine collection for testing, electrocardiogram (ECG) assessments (a measurement of the electrical activity of your heart), participant questionnaires, and physical examinations. TMC435 will be taken as an oral capsule of 150 mg once per day. Peginterferon (Pegasys ®) will be given as an injection of 180 µg once each week. Peginterferon (PegIntron®) will be given as an injection once each week and the dose will depend on your body weight. Ribavirin will be taken as a tablet (Copegus ®) or a capsule (Rebetol ®) twice each day and the dose will depend on your body weight.

ELIGIBILITY:
Inclusion Criteria:

* Genotype 1 hepatitis C infection (confirmed at screening)
* Participant has not received any prior treatment for hepatitis C
* Participant must have had a liver biopsy within 3 years before screening (or between the screening and baseline visit) showing chronic hepatitis C infection
* Must agree to use 2 forms of effective contraception throughout study (both males and females)

Exclusion Criteria:

* Infection with HIV or non genotype 1 hepatitis C
* Liver disease not related to hepatitic C infection
* Hepatic decompensation
* Significant laboratory abnormalities or other active diseases
* Pregnant or planning to become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 393 (Actual)
Dates: Start 2011-03; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen R&D Ireland Clinical Trial, Study Director — Janssen R&D Ireland
Locations (60):
- United States (11):
  - Los Angeles, California
  - Jacksonville, Florida
  - Orlando, Florida
  - Atlanta, Georgia
  - Crestview Hills, Kentucky
  - New Orleans, Louisiana
  - Saint Paul, Minnesota
  - Germantown, Tennessee
  - Houston, Texas
  - San Antonio, Texas
  - Falls Church, Virginia
- Argentina (2):
  - Buenos Aires
  - Rosario, Santa Fe
- Vienna, Austria
- Belgium (5):
  - Antwerp
  - Bruges
  - Brussels
  - Ghent
  - Leuven
- Brazil (2):
  - Salvador
  - São Paulo
- Bulgaria (2):
  - Plovdiv
  - Sofia
- France (5):
  - Clichy
  - Créteil
  - Nice
  - Paris
  - Vandœuvre-lès-Nancy
- Germany (10):
  - Berlin
  - Düsseldorf
  - Freiburg im Breisgau
  - Halle
  - Hanover
  - Kiel
  - Leipzig
  - München
  - Münster
  - Ulm
- Netherlands (2):
  - Amsterdam-Zuidoost
  - Leiden
- Poland (7):
  - Bialystok
  - Bydgoszcz
  - Chorzów
  - Czeladź
  - Kielce
  - Krakow
  - Warsaw
- Portugal (3):
  - Coimbra
  - Lisbon
  - Porto
- Santurce, Puerto Rico
- Slovakia (2):
  - Bratislava
  - Martin
- Spain (4):
  - Barcelona
  - Madrid
  - Seville
  - Valencia
- Turkey (Türkiye) (3):
  - Ankara
  - Istanbul
  - Izmir

REFERENCES:
- [Derived] Lenz O, Verbinnen T, Fevery B, Tambuyzer L, Vijgen L, Peeters M, Buelens A, Ceulemans H, Beumont M, Picchio G, De Meyer S. Virology analyses of HCV isolates from genotype 1-infected patients treated with simeprevir plus peginterferon/ribavirin in Phase IIb/III studies. J Hepatol. 2015 May;62(5):1008-14. doi: 10.1016/j.jhep.2014.11.032. Epub 2014 Nov 28. PMID 25445400
- [Derived] Manns M, Marcellin P, Poordad F, de Araujo ES, Buti M, Horsmans Y, Janczewska E, Villamil F, Scott J, Peeters M, Lenz O, Ouwerkerk-Mahadevan S, De La Rosa G, Kalmeijer R, Sinha R, Beumont-Mauviel M. Simeprevir with pegylated interferon alfa 2a or 2b plus ribavirin in treatment-naive patients with chronic hepatitis C virus genotype 1 infection (QUEST-2): a randomised, double-blind, placebo-controlled phase 3 trial. Lancet. 2014 Aug 2;384(9941):414-26. doi: 10.1016/S0140-6736(14)60538-9. Epub 2014 Jun 4. PMID 24907224

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted from 18 January 2011 to 5 February 2013. The study was conducted at 76 sites in 14 countries.
Pre-assignment Details: 393 participants were randomly allocated to the 2 treatment arms. 391 participants received at least 1 dose of study medication and were included in the intent-to-treat analysis set.
Groups:
- TMC435 150mg 12Wks PR24/48: Participants were given TMC435 150 mg once daily plus peginterferon alpha-2a/b (PegIFN alpha-2a/b) and ribavirin (RBV) for 12 Weeks (Wks) followed by PegIFN alpha-2a/b (P) and RBV (R) until Week 24 (PR24). Treatment was to be stopped at Week 24 for participants who achieved HCV RNA < 25 IU/mL detectable or undetectable at Week 4 and undetectable HCV RNA at Week 12. Other participants continued PR until Week 48 (PR48).
- PBO 12Wks PR48: Participants were given placebo (PBO) once daily plus peginterferon alpha-2a/b (PegIFN alpha-2a/b) and ribavirin (RBV) for 12 Weeks (Wks) followed by PegIFN alpha-2a/b (P) and RBV (R) until Week 48 (PR 48).
Period: Overall Study
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Started | 257 (Not including 1 participant was randomized to this group, but never received treatment.) | 134 (Not including 1 participant was randomized to this group, but never received treatment.)
Completed | 241 | 113
Not Completed | 16 | 21
Not completed — Adverse Event | 2 | 0
Not completed — Lost to Follow-up | 8 | 10
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 6 | 5
Not completed — Subject Entered Another Trial | 0 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48 | Total
Number analyzed (Participants) | 257 | 134 | 391
Age, Continuous [Median (Full Range); unit: years] | 46 [18 to 73] | 47 [18 to 73] | 47 [18 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 117 | 57 | 174
  Male | 140 | 77 | 217

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Participants Achieving a Sustained Virologic Response 12 Weeks After the Planned End of Treatment (SVR12)
Description: The table below shows the percentage of participants in each treatment group who achieved a SVR12, defined as the percentage of participants with undetectable plasma Hepatitis C virus ribonucleic acid 12 weeks after planned end of treatment.
Time Frame: Week 36 or Week 60
Population: The intent-to-treat population (defined as all participants who were randomized and received at least one dose of study medication) was used for all analyses.
Measure: Number; unit: Percentage of participants
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 257 | 134
Percentage of participants | 81.3 | 50.0
Statistical Analysis 1: Comparison: TMC435 150mg 12Wks PR24/48 vs PBO 12Wks PR48; The null hypothesis is there is no difference in proportions of SVR12 between the treatment groups; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Difference in proportions of SVR12 = 32.2, 95% CI 2-sided [23.3 to 41.2]

2. Secondary Outcome: The Percentage of Participants Achieving a Sustained Virologic Response at Week 72 (SVRW72)
Description: The table below shows the percentage of participants in each treatment group who achieved a SVRW72, defined as the percentage of participants with undetectable plasma Hepatitis C virus ribonucleic acid levels at end of treatment (EOT) and at Week 72.
Time Frame: Week 72
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 257 | 134
Percentage of participants | 78.6 | 50.0
Statistical Analysis 1: Comparison: TMC435 150mg 12Wks PR24/48 vs PBO 12Wks PR48; The null hypothesis is there is no difference in proportions of SVRW72 between the treatment groups; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Difference in proportions of SVRW72 = 29.3, 95% CI 2-sided [20.2 to 38.5]

3. Secondary Outcome: The Percentage of Participants Who Achieved a Sustained Virologic Response 24 Weeks After the Planned End of Treatment (SVR24)
Description: The table below shows the percentage of participants in each treatment group who achieved a SVR24, defined as the percentage of participants with undetectable plasma Hepatitis C virus ribonucleic acid levels 24 weeks after planned end of treatment.
Time Frame: Week 48 or Week 72
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 257 | 134
Percentage of participants | 80.5 | 50.0
Statistical Analysis 1: Comparison: TMC435 150mg 12Wks PR24/48 vs PBO 12Wks PR48; The null hypothesis is there is no difference in proportions of SVR24 between the treatment groups; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Difference in proportions of SVR24 = 31.5, 95% CI 2-sided [22.5 to 40.5]

4. Secondary Outcome: The Percentage of Participants Who Achieved a Sustained Virologic Response 4 Weeks After the Planned End of Treatment (SVR4)
Description: The table below shows the percentage of participants in each treatment group who achieved a SVR4, defined as the percentage of participants with undetectable plasma Hepatitis C virus ribonucleic acid levels 4 weeks after planned end of treatment.
Time Frame: Week 28 or Week 52
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 257 | 134
Percentage of participants | 84.8 | 53.0
Statistical Analysis 1: Comparison: TMC435 150mg 12Wks PR24/48 vs PBO 12Wks PR48; The null hypothesis is there is no difference in proportions of SVR4 between the treatment groups; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Difference in proportions of SVR4 = 32.3, 95% CI 2-sided [23.5 to 41.0]

5. Secondary Outcome: Change From Baseline in log10 Hepatitis C Virus (HCV) Ribonucleic Acid (RNA)
Description: The table below shows changes from baseline in log10 HCV RNA.
Time Frame: Day 3, Week 1, Week 4, Week 12, Week 24, and Week 48
Population: as for outcome 1
Measure: Mean (Standard Error); unit: log10 IU/mL
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 257 | 134
log10 IU/mL
  Day 3 | -3.60 (0.045) | -1.22 (0.075)
  Week 1 | -4.52 (0.043) | -1.21 (0.094)
  Week 4 | -5.28 (0.046) | -2.72 (0.138)
  Week 12 | -5.34 (0.053) | -4.21 (0.129)
  Week 24 | -5.27 (0.062) | -4.93 (0.114)
  Week 48 | -5.83 (0.074) | -5.28 (0.084)

6. Secondary Outcome: Actual Values of log10 Hepatitis C Virus (HCV) Ribonucleic Acid (RNA)
Description: The table below shows actual values of log10 HCV RNA levels.
Time Frame: Day 3, Week 1, Week 4, Week 12, Week 24, and Week 48
Population: as for outcome 1
Measure: Mean (Standard Error); unit: log10 IU/mL
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 257 | 134
log10 IU/mL
  Day 3 | 2.777 (0.050) | 5.165 (0.107)
  Week 1 | 1.852 (0.400) | 5.171 (0.129)
  Week 4 | 1.093 (0.027) | 3.657 (0.162)
  Week 12 | 1.027 (0.034) | 2.157 (0.141)
  Week 24 | 1.094 (0.049) | 1.388 (0.106)
  Week 48 | 1.015 (0.061) | 0.960 (0.005)

7. Secondary Outcome: Percentage of Participants With On-treatment Virologic Response at All Time Points
Description: The table below shows the percentage of participants with Hepatitis C Virus (HCV) ribonucleic acid (RNA) plasma levels below the limit of detection (ie, <25 IU/mL undetectable), the percentage of participants with a HCV RNA plasma level below the limit of quantification (ie, less than [<] 25 IU/mL detectable or undetectable), the percentage of participants with plasma levels of HCV RNA <100 IU/mL, the percentage of HCV-Infected participants with virologic responses of a greater than or equal to 2 log10 change from baseline in plasma levels of HCV RNA.
Time Frame: Day 3, Week 1, Week 2, Week 8, Week 16, Week 20, Week 28, Week 36, and Week 42
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 257 | 134
Percentage of participants
  Day 3:<25 IU/mL undetectable | 0.4 | 0
  Week 1:<25 IU/mL undetectable | 6.3 | 1.5
  Week 2:<25 IU/mL undetectable | 31.7 | 3.8
  Week 8:<25 IU/mL undetectable | 93.7 | 31.3
  Week 16:<25 IU/mL undetectable | 96.3 | 65.5
  Week 20:<25 IU/mL undetectable | 95.9 | 68.2
  Week 28:<25 IU/mL undetectable | 66.7 | 88.0
  Week 36:<25 IU/mL undetectable | 100.0 | 95.3
  Week 42:<25 IU/mL undetectable | 100.0 | 95.0
  Day 3:<25 IU/mL detectable or undetectable | 4.7 | 0
  Week 1:<25 IU/mL detectable or undetectable | 37.0 | 2.3
  Week 2:<25 IU/mL detectable or undetectable | 80.7 | 12.0
  Week 8:<25 IU/mL detectable or undetectable | 98.0 | 45.0
  Week 16:<25 IU/mL detectable or undetectable | 98.0 | 73.5
  Week 20:<25 IU/mL detectable or undetectable | 97.1 | 79.1
  Week 28:<25 IU/mL detectable or undetectable | 77.8 | 97.8
  Week 36:<25 IU/mL detectable or undetectable | 100.0 | 98.8
  Week 42:<25 IU/mL detectable or undetectable | 100.0 | 100.0
  Day 3:<100 IU/mL | 15.3 | 1.5
  Week 1:<100 IU/mL | 65.7 | 6.0
  Week 2:<100 IU/mL | 92.0 | 14.3
  Week 8:<100 IU/mL | 98.8 | 50.4
  Week 16:<100 IU/mL | 98.8 | 77.0
  Week 20:<100 IU/mL | 98.0 | 83.6
  Week 28:<100 IU/mL | 77.8 | 97.8
  Week 36:<100 IU/mL | 100.0 | 98.8
  Week 42:<100 IU/mL | 100.0 | 100.0
  Day 3:> or = 2 log 10 change from baseline | 96.9 | 20.8
  Week 1:> or =2 log 10 change from baseline | 99.6 | 24.1
  Week 2:> or =2 log 10 change from baseline | 99.6 | 39.8
  Week 8:> or =2 log 10 change from baseline | 99.6 | 80.2
  Week 16:> or =2 log 10 change from baseline | 99.2 | 97.3
  Week 20:> or =2 log 10 change from baseline | 98.8 | 93.6
  Week 28:> or =2 log 10 change from baseline | 88.9 | 100.0
  Week 36:> or =2 log 10 change from baseline | 100.0 | 98.8
  Week 42:> or =2 log 10 change from baseline | 100.0 | 100.0

8. Secondary Outcome: The Percentage of Participants Achieving a Rapid Virologic Response (RVR)
Description: The table below shows the percentage of participants in each treatment group who achieved a RVR, defined as having undetectable plasma Hepatitis C virus ribonucleic acid levels after receiving 4 weeks of treatment.
Time Frame: Week 4
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 257 | 134
Percentage of participants | 79.2 | 12.8

9. Secondary Outcome: The Percentage of Participants Achieving a Early Virologic Response (EVR)
Description: The table below shows the percentage of participants who achieved an EVR, defined as having a change from baseline in plasma Hepatitis C virus ribonucleic acid of 2 log10 at Week 12.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 257 | 134
Percentage of participants | 98.8 | 89.8

10. Secondary Outcome: The Percentage of Participants Achieving a Complete Early Virologic Response (cEVR)
Description: The table below shows the percentage of participants in each treatment group who had a cEVR, defined as having undetectable plasma Hepatitis C Virus ribonucleic acid levels at Week 12.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 257 | 134
Percentage of participants | 96.8 | 44.9

11. Secondary Outcome: The Percentage of Participants Achieving a Extended Rapid Virologic Response (eRVR)
Description: The table below shows the percentage of participants in each treatment group who had a eRVR, defined as having undetectable plasma Hepatitis C Virus ribonucleic acid levels at Week 4 and 12.
Time Frame: Weeks 4 and 12
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 257 | 134
Percentage of participants | 78.3 | 13.4

12. Secondary Outcome: The Percentage of Participants With <1 log10 Decrease in Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) From Baseline at Week 4
Description: The table below shows the percentage of participants in each treatment group with <1 log10 HCV RNA decrease at Week 4.
Time Frame: Week 4
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 257 | 134
Percentage of participants | 0.4 | 17.3

13. Secondary Outcome: Percentage of Participants With in Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) Levels >1000 IU/mL at Week 4
Description: The table below shows the percentage of participants in each treatment group with HCV RNA levels >1000 IU/mL at Week 4.
Time Frame: Week 4
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 257 | 134
Percentage of participants | 1.2 | 61.2

14. Secondary Outcome: Percentage of Participants With Null Response
Description: The table below shows the percentage of participants with null response, defined as <2 log10 reduction in Hepatitis C virus ribonucleic acid at Week 12 compared to baseline.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 257 | 134
Percentage of participants | 1.2 | 10.2

15. Secondary Outcome: Percentage of Participants With Partial Response
Description: The table below shows the percentage of participants with partial response, defined as =>2 log10 reduction in Hepatitis C virus (HCV) ribonucleic acid (RNA) at Week 12 compared to baseline, but not achieving undetectable HCV RNA while on treatment.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 257 | 134
Percentage of participants | 0.4 | 17.3

16. Secondary Outcome: Percentage of Participants With Viral Breakthrough
Description: The table below shows the percentage of participants with viral breakthrough, defined as a confirmed increase of greater than 1 log10 IU/mL in plasma Hepatitis C virus (HCV) ribonucleic acid (RNA) level from the lowest level reached (ie, lowest value measured in between baseline and current value), or a confirmed plasma HCV RNA level of greater than 100 IU/mL in participants whose plasma HCV RNA had previously been below the limit of quantification (25 IU/mL detectable) or undetectable (<25 IU/mL undetectable).
Time Frame: Up to Week 48
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 257 | 134
Percentage of participants | 4.7 | 10.4

17. Secondary Outcome: Percentage of Participants With Viral Relapse
Description: The table below shows the percentage of participants with viral relapse, defined as having confirmed detectable plasma level of Hepatitis C virus (HCV) ribonucleic acid (RNA) during the follow-up period in participants with undetectable plasma HCV RNA (<25 IU/mL undetectable) at the end of treatment.
Time Frame: Up to Week 72
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 257 | 134
Percentage of participants | 12.3 | 23.9

18. Secondary Outcome: Percentage of Participants Who Completed All Study Treatment at Week 24 Because of the Treatment Duration Rule
Description: The table below shows the percentage of participants in the TMC435 treatment group who met the treatment duration rule (ie, having hepatitis C virus [HCV] ribonucleic acid [RNA] levels <25 IU/mL detectable or undetectable at Week 4 and undetectable HCV RNA levels at Week 12) and completed treatment with PegIFNα-2a and RBV for 24 weeks. Participants in the TMC435 treatment group not meeting RGT criteria and participants in the placebo group were treated with PegIFNα-2a and RBV treatment for 48 weeks.
Time Frame: Week 24
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 257 | 134
Percentage of participants | 89.5 | NA — RGT criteria did not apply to PBO arm

19. Secondary Outcome: Percentage of Participants With On-treatment Failure
Description: The table below shows percentage of participants with on-treatment failure defined as confirmed detectable Hepatitis C virus ribonucleic acid levels at actual end of treatment.
Time Frame: Week 48
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 257 | 134
Percentage of participants | 7.0 | 32.1

20. Secondary Outcome: Time to Reach Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) <25 IU/mL Undetectable or Detectable
Description: The table below shows the median time in days to reach HCV RNA levels <25 IU/mL undetectable or detectable.
Time Frame: Up to Week 48
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 257 | 134
Days | 14 [14 to 15] | 85 [57 to 112]

21. Secondary Outcome: Time to Reach Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) <25 IU/mL Undetectable
Description: The table below shows the median time in days to reach HCV RNA levels <25 IU/mL undetectable.
Time Frame: Up to Week 48
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 257 | 134
Days | 29 [28 to 29] | 113 [85 to 141]

22. Secondary Outcome: Time to Reach Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) <100 IU/mL
Description: The table below shows the median time in days to reach HCV RNA levels <100 IU/mL.
Time Frame: Up to Week 48
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 257 | 134
Days | 8 [NA to NA] — The 95% CI could not be calculated due to very low number of failures in the TMC435 group. | 71 [57 to 86]

23. Secondary Outcome: Time to Reach Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) <1000 IU/mL
Description: The table below shows the median time in days to reach HCV RNA levels <1000 IU/mL.
Time Frame: Up to Week 48
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 257 | 134
Days | 4 [3 to 4] | 57 [56 to 58]

24. Secondary Outcome: The Percentage of Participants With Viral Breakthrough at Different Time Points
Description: The table below shows the percentage of participants at different time points with viral breakthrough, defined as a confirmed increase of greater than 1 log10 IU/mL in plasma HCV ribonucleic acid (RNA) level from the lowest level reached (ie, lowest value measured in between baseline and current value), or a confirmed plasma HCV RNA level of greater than 100 IU/mL in participants whose plasma HCV RNA had previously been below the limit of quantification (25 IU/mL detectable) or undetectable (<25 IU/mL undetectable).
Time Frame: Up to Week 48
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 257 | 134
Percentage of participants
  < 12 Weeks | 1.2 | 3.7
  Week 12 - Week 24 | 3.3 | 6.4
  > Week 24 | 12.5 | 2.1

25. Secondary Outcome: Time From End-of-treatment to Viral Relapse
Description: The table below shows the mean number of days to viral relapse, defined as participants having confirmed detectable plasma level of Hepatitis C Virus (HCV) ribonucleic acid (RNA) during the follow-up period in participants with undetectable plasma HCV RNA (<25 IU/mL undetectable) at the end of treatment.
Time Frame: Up to Week 72
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Days
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 257 | 134
Days | 229.77 (4.29) | 77.74 (2.34)

26. Secondary Outcome: The Percentage of Participants With Normalization of Alanine Aminotransferase (ALT)
Description: The percentage of participants analyzed were those with baseline ALT values out of the normal range (ie, 164 of 257 participants in the TMC435 treatment group and 79 of 134 participants in the Placebo group had ALT values at baseline that were out of the normal range.). Normalization of ALT values means that ALT values out of the normal range returned to within the normal range.
Time Frame: Up to Week 48
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 169 | 79
Percentage of participants | 79.9 | 81.0

27. Secondary Outcome: Median Time to Normalization of Alanine Aminotransferase (ALT) Levels
Description: The table below shows the median time in weeks to normalization of ALT levels.
Time Frame: Up to Week 48
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 257 | 134
Weeks | 2.14 [1.29 to 2.14] | 4.14 [4.14 to 12.00]

28. Secondary Outcome: Plasma Concentration of TMC435: Area Under the Plasma Concentration-time Curve From the Time of Administration to 24 Hours After Dosing (AUC24h)
Description: The table below shows the mean (standard deviation) values of the area under the plasma concentration-time curve from time of administration to 24 hours after dosing for TMC435.
Time Frame: At protocol-specified time points from the time of administration up to 24 hours after dosing at Weeks 2, 4, 8, and 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | TMC435 150mg 12Wks PR24/48
Number analyzed (Participants) | 255
ng*h/mL | 56611 (66935.4)

29. Secondary Outcome: Plasma Concentration of TMC435: Predose Plasma Concentration (C0h)
Description: The table below shows the mean (standard deviation) of C0h values of TMC435. NOTE: the timing of collection of blood samples post-dose for analysis at Week 2, 4, 8, and 12 was not specifed; only the interval was between blood samples was specified (ie, 2 samples collected 2 hours apart at Week 2, 4, 8, and 12).
Time Frame: Blood samples tested were taken before administration of TMC435 and at 2 random time points after dosing (taken atleast 2 hours apart from each other) at Week 2, 4, 8, and 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | TMC435 150mg 12Wks PR24/48
Number analyzed (Participants) | 255
ng/mL | 1902 (2781.1)

30. Secondary Outcome: Plasma Concentration of TMC435: Systemic Clearance (CL)
Description: The table below shows the mean (standard deviation) of CL values of TMC435. NOTE: the pre-dose CL values taken at Weeks, 2, 4, 8, and 12 were averaged and then the mean values from all participants were averaged to provide the final value reported below.
Time Frame: At protocol-specified time points at Weeks 2, 4, 8, and 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | TMC435 150mg 12Wks PR24/48
Number analyzed (Participants) | 255
L/h | 5.23 (3.767)

31. Secondary Outcome: Area Under the Curve From Baseline to Week 60 (AUC60) and Week 72 (AUC72) for the Fatigue Severity Scale (FSS) Total Scores
Description: Study participants completed FSS questionnaires during study visits before treatment and throughout follow-up to rate the severity and impact of fatigue experienced in the preceding 2 weeks. FSS total scores are the average of nine questions with a range from 1 [no fatigue] to 7 [worst fatigue]; the possible score range from baseline to Week 60 would be 60-420 and to Week 72 would be 72-504. The average FSS total score from baseline to Week 60 and to Week 72 was calculated for each participant and then the average of those values were calculated to show the average FSS total score for each treatment group. The null hypothesis was that there would be no difference between the treatment arms in the FSS total score. The Table below shows the lease squares (LS) mean estimates of the area under the curve (AUC) at Week 72 (as well as at Week 60) and the statistical comparison between treatment groups.
Time Frame: Baseline to Week 60 and Week 72
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale*weeks
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 256 | 133
Scores on a scale*weeks
  Week 60 | 208.418 [199.4881 to 217.3476] | 225.194 [213.8370 to 236.5513]
  Week 72 | 240.695 [230.1386 to 251.2542] | 259.532 [246.0810 to 272.9834]
Statistical Analysis 1: Comparison: TMC435 150mg 12Wks PR24/48 vs PBO 12Wks PR48; Fatigue Severity Score AUC60; Test type: Superiority or Other; p = 0.008, Piecewise Linear Model; Mean differences = -16.776, 95% CI 2-sided [-29.1502 to -4.4025], Standard Error of Mean 6.3081
Statistical Analysis 2: Comparison: TMC435 150mg 12Wks PR24/48 vs PBO 12Wks PR48; Fatigue Severity Score AUC72; Test type: Superiority or Other; p = 0.012, Piecewise Linear Model; Mean differences = -18.837, 95% CI 2-sided [-33.4933 to -4.1801], Standard Error of Mean 7.4715

32. Secondary Outcome: Area Under the Curve From Baseline to Week 60 (AUC60) and Week 72 (AUC72) for Impairment in Overall Work Productivity Due to Hepatitis C Virus (HCV) Infection and Its Treatment
Description: Impairment in overall work productivity was measured using the Work Productivity and Activity Impairment (WPAI): Hepatitis C questionnaire completed by participants throughout the study. WPAI Overall Productivity Scores ranged from 0% to 100% (higher WPAI scores indicated greater impairment in productivity). The average WPAI score from baseline to Week 72 was calculated for each participant and then the average of those values were calculated to show the average WPAI score for each treatment group. The null hypothesis was there is no statistically significant difference between the treatment groups in the AUC for the change from baseline to Week 72 (AUC72) in WPAI Productivity Scores. The Table below shows WPAI Productivity Scores at Week 72 (as well as at Week 60) from the model used to calculate the AUC and the statistical comparison between treatment groups.
Time Frame: Baseline to Week 60 and Week 72
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale*weeks
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 256 | 133
Scores on a scale*weeks
  Week 60 | 1628.075 [1492.3021 to 1763.8485] | 1910.235 [1730.5026 to 2089.9681]
  Week 72 | 1781.768 [1622.4802 to 1941.0560] | 2106.131 [1894.8814 to 2317.3811]
Statistical Analysis 1: Comparison: TMC435 150mg 12Wks PR24/48 vs PBO 12Wks PR48; Impairment in Work Productivity AUC60; Test type: Superiority or Other; p = 0.008, Piecewise Linear Model; Mean differences = -282.160, 95% CI 2-sided [-489.1252 to -75.1949], Standard Error of Mean 105.4927
Statistical Analysis 2: Comparison: TMC435 150mg 12Wks PR24/48 vs PBO 12Wks PR48; Impairment in Work Productivity AUC72; Test type: Superiority or Other; p = 0.009, Piecewise Linear Model; Mean differences = -324.363, 95% CI 2-sided [-567.7080 to -81.0182], Standard Error of Mean 124.0260

33. Secondary Outcome: Area Under the Curve From Baseline to Week 60 (AUC60) and Week 72 (AUC72) for Impairment in Daily Activities Due to Hepatitis C Virus (HCV) Infection and Its Treatment
Description: Impairment in daily activity was measured using the Work Productivity and Activity Impairment (WPAI): Hepatitis C questionnaire, Question 6. The possible impairment in WPAI daily activity score range from baseline to Week 60 was 0-6000 and to Week 72 was 0-7200, with the higher scores indicating more impairment in daily activities. The average WPAI impairment in daily activity score from baseline to Week 72 was calculated for each participant and then the average of those values were calculated to show the average WPAI impairment in daily activity score for each treatment group. The null hypothesis was there is no statistically significant difference between the treatment arms in the AUC for the change from baseline to Week 72 (AUC72) in WPAI impairment in daily activity scores. The Table below shows the WPAI Impairment in daily activity scores at Week 72 (as well as at Week 60) and the statistical analysis between treatment groups.
Time Frame: Baseline to Week 60 and Week 72
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale*weeks
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 256 | 133
Scores on a scale*weeks
  Week 60 | 1580.635 [1445.8307 to 1715.4397] | 1863.071 [1684.4355 to 2041.7065]
  Week 72 | 1727.079 [1568.9831 to 1885.1745] | 2056.283 [1846.3791 to 2266.1868]
Statistical Analysis 1: Comparison: TMC435 150mg 12Wks PR24/48 vs PBO 12Wks PR48; Impairment in Daily Activities AUC60; Test type: Superiority or Other; p = 0.007, Piecewise linear model; Mean Differences = -282.436, 95% CI 2-sided [-488.4150 to -76.4566], Standard Error of Mean 104.9894
Statistical Analysis 2: Comparison: TMC435 150mg 12Wks PR24/48 vs PBO 12Wks PR48; Impairment in Daily Activities AUC72; Test type: Superiority or Other; p = 0.008, Piecewise Linear Model; Mean differences = -329.204, 95% CI 2-sided [-571.3389 to -87.0695], Standard Error of Mean 123.4080

34. Secondary Outcome: Area Under the Curve From Baseline to Week 60 (AUC60) and Week 72 (AUC72) for Time Missed From Work Due to Hepatitis C Virus (HCV) Infection and Its Treatment
Description: Hours missed from work because of HCV infection or its treatment was assessed by measuring the change from baseline in the Work Productivity and Activity Impairment (WPAI): Hepatitis C questionnaire Absenteeism score (time missed from work). The possible WPAI WPAI absenteeism score range from baseline to Week 60 was 0-6000 and to Week 72 was 0-7200, with the higher scores indicating more impairment in WPAI absenteeism. The average WPAI absenteeism score from baseline to Week 60/72 was calculated for each participant and then the average of those values calculated for each treatment group. The area under the curve (AUC60/AUC72) over time from baseline to Week 60/72 was derived from a piecewise-linear model allowing the slopes to change at Week 4, 12, 24, 36, 48 and 60. The null hypothesis was there is no statistically significant difference between the treatment arms in the area under the curve (AUC) from baseline to Week 72 (AUC72) in WPAI absenteeism score.
Time Frame: Baseline to Week 60 and Week 72
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale*weeks
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 182 | 89
Scores on a scale*weeks
  Week 60 | 653.642 [511.4925 to 795.7918] | 840.495 [637.5293 to 1043.4599]
  Week 72 | 698.223 [533.6236 to 862.8224] | 886.425 [650.2224 to 1122.6266]
Statistical Analysis 1: Comparison: TMC435 150mg 12Wks PR24/48 vs PBO 12Wks PR48; Time Missed from Work AUC60; Test type: Superiority or Other; p = 0.125, Piecewise linear model; Mean differences = -186.852, 95% CI 2-sided [-425.4109 to 51.7059], Standard Error of Mean 121.4741
Statistical Analysis 2: Comparison: TMC435 150mg 12Wks PR24/48 vs PBO 12Wks PR48; Time Missed from Work AUC72; Test type: Superiority or Other; p = 0.183, Piecewise linear model; Mean differences = -188.202, 95% CI 2-sided [-465.5070 to 89.1040], Standard Error of Mean 141.1702

ADVERSE EVENTS:
Time Frame: 72 weeks
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Serious Adverse Events (participants affected / at risk) | 16/257 | 10/134
Other Adverse Events (participants affected / at risk) | 243/257 | 131/134
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TMC435 150mg 12Wks PR24/48 (N=257) | PBO 12Wks PR48 (N=134)
Anal abscess (Infections and infestations) | 1 | 0
Lymphadenitis bacterial (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 0 | 1
Epilepsy (Nervous system disorders) | 1 | 0
Memory impairment (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 1
Thoracic outlet syndrome (Nervous system disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 2 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Hyphaema (Eye disorders) | 1 | 0
Visual impairment (Eye disorders) | 1 | 0
Retinal ischaemia (Eye disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Mixed deafness (Ear and labyrinth disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0
Enterocutaneous fistula (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Death (General disorders) | 1 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Aggression (Psychiatric disorders) | 1 | 0
Drug abuse (Psychiatric disorders) | 0 | 1
Angina unstable (Cardiac disorders) | 0 | 1
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TMC435 150mg 12Wks PR24/48 (N=257) | PBO 12Wks PR48 (N=134)
Fatigue (General disorders) | 95 | 56
Pyrexia (General disorders) | 80 | 53
Influenza like illness (General disorders) | 66 | 35
Asthenia (General disorders) | 59 | 38
Chills (General disorders) | 21 | 12
Injection site erythema (General disorders) | 15 | 9
Pruritus (Skin and subcutaneous tissue disorders) | 65 | 34
Rash (Skin and subcutaneous tissue disorders) | 46 | 15
Alopecia (Skin and subcutaneous tissue disorders) | 43 | 27
Dry skin (Skin and subcutaneous tissue disorders) | 28 | 18
Eczema (Skin and subcutaneous tissue disorders) | 4 | 9
Headache (Nervous system disorders) | 101 | 49
Dizziness (Nervous system disorders) | 21 | 9
Disturbance in attention (Nervous system disorders) | 13 | 8
Dysgeusia (Nervous system disorders) | 6 | 7
Nausea (Gastrointestinal disorders) | 63 | 24
Diarrhoea (Gastrointestinal disorders) | 34 | 12
Vomiting (Gastrointestinal disorders) | 17 | 7
Dry mouth (Gastrointestinal disorders) | 13 | 6
Abdominal pain (Gastrointestinal disorders) | 12 | 7
Abdominal pain upper (Gastrointestinal disorders) | 11 | 12
Constipation (Gastrointestinal disorders) | 8 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 58 | 28
Arthralgia (Musculoskeletal and connective tissue disorders) | 32 | 14
Back pain (Musculoskeletal and connective tissue disorders) | 25 | 13
Muscle spasms (Musculoskeletal and connective tissue disorders) | 8 | 7
Insomnia (Psychiatric disorders) | 51 | 21
Depression (Psychiatric disorders) | 29 | 19
Mood altered (Psychiatric disorders) | 22 | 15
Anxiety (Psychiatric disorders) | 17 | 6
Sleep disorder (Psychiatric disorders) | 13 | 5
Neutropenia (Blood and lymphatic system disorders) | 49 | 29
Anaemia (Blood and lymphatic system disorders) | 46 | 33
Thrombocytopenia (Blood and lymphatic system disorders) | 13 | 9
Leukopenia (Blood and lymphatic system disorders) | 10 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 32 | 22
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 23 | 11
Decreased appetite (Metabolism and nutrition disorders) | 46 | 21
Weight decreased (Investigations) | 14 | 6
Neutrophil count decreased (Investigations) | 8 | 7
Influenza (Infections and infestations) | 5 | 8
Sinusitis (Infections and infestations) | 5 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days